CLINICAL TRIAL: NCT05107024
Title: Resting Full-cycle Ratio-guided Step by Step Dilation for Drug-coated Balloon Treatment of de Novo Coronary Lesions (REDUCE) Study
Brief Title: Resting Full-cycle Ratio-guided Step by Step Balloon Dilation
Acronym: REDUCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shenzhen REDUCE
Record Dates: First submitted 2021-10-27; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: de Novo Coronary Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional balloon dilation group (Active Comparator): The optimal size of the semi-compliant balloon (balloon to vessel ratio 1.0) was determined by the surgeon according to angiography, and sufficient predilation was performed to achieve residual stenosis. 30% vascular anatomy criteria, and then a 1:1 DCB was selected for drug release
  Interventions: Device: Traditional balloon dilation
- RFR-guided step by step balloon dilation group (Experimental): Balloon dilation start with 2.0mm compliant balloon. After 8atm pressure expansion, the RFR value was measured. If RFR≥0.93, the pre-expansion was stopped. Otherwise, RFR value is measured after pressure expansion of 16atm, if RFR value is still less than 0.93, then a 2.5mm compliant or non-compliant balloon was used to expand the pressure of 8ATM, and the balloon diameter and expansion pressure were continuously increased until RFR≥0.93. Then a DCB with the same diameter as the pre-expanded balloon was selected for drug release.
  Interventions: Device: RFR-guided step by step balloon dilation

INTERVENTIONS:
Device: RFR-guided step by step balloon dilation — The mean value of the minimum ratio of distal mean pressure to aortic mean pressure (Pd/Pa) in five consecutive complete cardiac cycles was obtained by scanning the diastolic and systolic stages at rest.
  Arms: RFR-guided step by step balloon dilation group
Device: Traditional balloon dilation — The surgeon determines the optimal size of the semi-compliant balloon based on angiography (balloon to vessel ratio 1.0) and performs adequate predilation to achieve residual stenosis. 30% of vascular anatomy criteria
  Arms: Traditional balloon dilation group

SUMMARY:
Drug-coated balloon (DCB), as an implant-free treatment technique, has been widely used in coronary interventional therapy, effectively solving the problem of restenosis caused by traditional stent implantation, and providing a treatment option for patients with coronary heart disease with high blood risk. However, in DCB treatment of coronary artery lesions, the incidence of dissection is as high as 10-20% when the balloon is predilated, which often requires salvage stent implantation, resulting in the treatment failure of DCB and bringing great hidden dangers to patients. The main reason was that excessive balloon predilation was caused by the standard of vascular anatomy (residual lumen stenosis less than 30%). The resting full cycle ratio (RFR) is a reliable method for determining the presence of functional ischemia in coronary artery lesions and enables immediate detection. We hypothesized that RFR-guided stepped-balloon dilation could reduce the incidence of dissection and increase the success rate of DCB treatment. Fifty patients who planned to receive DCB treatment were randomly divided into balloon dilation alone (n=25) and RFR-guided stepped-balloon dilation group (n=25). The primary endpoint was the success rate of DCB treatment. This study will provide a functional evaluation based balloon predilation method for DCB treatment, making DCB treatment for orthotopic coronary artery disease more safe and effective.

DETAILED DESCRIPTION:
To compare the application of pre-treated lesions with DCB in the treatment of coronary artery disease in situ between the simple balloon dilation group and rFR-guided stepped-balloon dilation group.

It was a single-center, open, prospective, randomized controlled study. Fifty patients with symptoms of myocardial ischemia or relevant evidence for DCB treatment of coronary artery disease in situ were enrolled and randomly divided into balloon dilation group alone (n=25) and rFR-guided step balloon dilation group (n=25).

In the balloon dilation group, the optimal size of the semi-compliant balloon was determined by the surgeon according to angiography (the ratio of balloon to blood vessel was 1.0), and full predilation was performed to achieve residual stenosis. 30% vascular anatomy criteria, and then a 1:1 DCB was selected for drug release; The step balloon expansion group guided by RFR expanded from 2.0mm compliant balloon. After 8atm pressure expansion, the RFR value was measured. If RFR≥0.93, the pre-expansion was stopped. 0.93, RFR value is measured after pressure expansion of 16atm, if RFR&lt is still; 0.93, then a 2.5mm compliant or non-compliant balloon was used to expand the pressure of 8ATM, and the balloon diameter and expansion pressure were continuously increased until RFR≥0.93, and then A DCB with the same diameter as the pre-expanded balloon was selected for drug release. If c-type or higher dissection or TIMI flow occurs & LT; Grade 3 patients were given salvage stents.

Collect patient history and improve clinical examination; The occurrence and classification of dissection, final pre-dilated balloon diameter, DCB diameter, incidence of salvage stent implantation, residual stenosis, operation time, and radiation dose were recorded intraoperatively. The incidence of revascularization and angina pectoris during hospitalization were recorded. Minimum lumen diameter and diameter stenosis rate were detected by coronary angiography 9 months after discharge. MACE events were observed 12 months after discharge.

With residual lumens stenosis less than 30% as the criteria the pure balloon pre expansion of coronary artery lesions in situ can result in up to 10-40% of the incidence of retrospective stenting, limits the DCB in coronary artery lesions in situ treatment, the application of quasi simple balloon expansion and pathological changes of RFR guiding ladder balloon expansion of pretreatment in the DCB treatment of coronary artery lesions, the application of in situ To verify that rFR-guided stepped-balloon dilation compared with balloon dilation alone can increase the success rate of DCB in the treatment of orthotopic coronary artery lesions, thus providing a new pre-dilation treatment method for DCB to be more effective and safe in the application of orthotopic coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old; Presenting with stable or unstable angina and/or evidence of myocardial ischemia; The treated lesions were in situ coronary artery lesions. Angiography showed lumen diameter of 2.5-4.0mm and diameter stenosis ≥80%. No more than 2 lesions require treatment.

Exclusion Criteria:

* Acute myocardial infarction within 48 hours of onset; Life expectancy of less than 12 months; Lesion in left main trunk, lesion length > 24mm, severe calcification, thrombosis or bifurcation; There are other lesions that require stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of DCB treatment | During sample collection (1 year)
  Successful DCB treatment was defined as the use of DCB-releasing agents in the treatment of orthotopic coronary artery disease without the need for salvage stent implantation during surgery and hospitalization

SECONDARY OUTCOMES:
Incidence of adverse cardiac events (MACE) | 2 years
  All-cause death, myocardial infarction, target vessel remodeling (TVR), and vascular thrombosis
Incidence of late lumen loss | 2 years
  Analysis of the minimum lumen diameter after operation and the minimum lumen diameter of the same vascular segment

CONTACTS AND LOCATIONS:
Overall Officials: Shaohong Dong, Study Chair — Shenzhen People's Hospital

IPD SHARING:
Plan to Share IPD: No